CLINICAL TRIAL: NCT02841436
Title: A Clinical Research About Using Irreversible Electroporation to Treat Locally Advanced Pancreatic Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201210008DIC
Record Dates: First submitted 2016-06-27; First posted 2016-07-22 (Estimated); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Pancreatic Cancer
Keywords: irreversible electroporation; pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Electroporation; Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- irreversible electroporation (IRE) (Experimental): IRE (AngioDynamics, NY) To use 2 to 6 unipolar electrodes in a predetermined grid pattern. 90 pulses of 2,000 - 3,000 V were applied with a pulse generator (AngioDynamics, NY) across the gap between the electrodes for 100 microseconds (0.1 msec) per each ablation.
  Interventions: Device: Irreversible Electroporation (IRE) System

INTERVENTIONS:
Device: Irreversible Electroporation (IRE) System

SUMMARY:
Pancreatic cancers is one the most important malignancies with highest mortality in the world. The prognosis of these patients is very poor. Although some patients with early-diagnosed disease could receive surgical intervention, a majority (70%to 80%) of patients present with locally advanced or metastatic status are inoperable. Patients in this late status usually are recommended to receive palliative bypass operation such as choledochojejunostomy and/or gastrojejunostomy and palliative radiotherapy for the pancreatic cancer. Radiofrequency ablation (RFA) used to be expected an alternative therapy. However, the main drawback of RFA is its side effect to damage adjacent structure such as bile duct, and the tumors located adjacent to vessels could not be ablated well.

DETAILED DESCRIPTION:
Irreversible electroporation (IRE), developed and manufactured by AngioDynamics US Ltd, can ablate tumor by fenestrating the cancer cell membrane by electric pulse. The anti-tumor effect does not result from thermotherapy, so is also not diminished by adjacent vessels. Several pre-clinical and clinical studies have already demonstrated IRE is a safe and effective treatment, and the adjacent tissue such as vessels and ductal structures will be spared. Recently, IRE had been used to treat pancreatic cancer successfully, and the safety is satisfactory. The system has been approved as safe by the European Union (EU) in 2008 and received Food and Drug Administration (FDA) approval in 2010. However, there are still few experiences in using IRE for tumor ablation in Taiwan. In this study, the investigators will perform IRE for inoperable patients with locally advanced pancreatic cancers. They will receive IRE during the operation of palliative bypass operation including choledochojejunostomy and/or gastrojejunostomy. The investigators will evaluate the potential side effect and ablate effect of tumors, and also follow-up the patients for 2 years to evaluate the overall survival. The investigators will appraisal the clinical feasibility and advantage of the system by this study.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following inclusion criteria to be eligible for this study:

1. Locally advanced pancreatic cancer is defined as per the 7th edition of the American Joint Committee on Cancer (AJCC) staging system for pancreatic cancer -described as arterial encasement of either the celiac axis or superior mesenteric artery or both.
2. Biliary tract or intestine is compromised by tumor, palliative bypass operation (hepaticojejunostomy and/or gastrojejunostomy) is considered to be performed.
3. Eastern Cooperative Oncology Group (ECOG) score of 0-1,
4. American Society of Anaesthesiologists (ASA) score ≤ 3,
5. Adequate bone marrow, liver and renal function. Platelet count ≥ 100 K/Μl. Total bilirubin ≦ 5 mg/dL. alanine transaminase (ALT) and aspartate transaminase (AST) < 5 x upper limit of normal. prothrombin time (PT)- international normalized ratio (INR) ≦ 2.0 (5). Serum creatinine ≦ 1.5 x upper limit of normal
6. Prior Informed Consent Form
7. Life expectancy of at least 3 months.

Exclusion Criteria:

Patients presenting with any of the following will not be enrolled into this study:

1. History of cardiac disease:
2. Congestive heart failure >New York Heart Association (NYHA) class 2
3. Active coronary artery disease (CAD) (myocardial infarction more than 6 months prior to study entry is allowed)
4. Cardiac arrhythmias (>Grade 2 NCI-CTCAE Version 3.0) which are poorly controlled with anti-arrhythmic therapy or requiring pace maker
5. Uncontrolled hypertension
6. Any active metal implanted device (eg Pacemaker),
7. Women who are pregnant or women of child-bearing potential who are not using an acceptable method of contraception,
8. Received treatment with an investigational agent/ procedure within 30 days prior to treatment with the IRE System,
9. Known history of human immunodeficiency virus (HIV) infection
10. Patients with resectable lesions.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2012-11; Primary Completion 2014-06-16 (Actual); Study Completion 2020-05-27 (Actual)

PRIMARY OUTCOMES:
Tumor response | 1 month after treatment
  Tumor response will be evaluated by abdominal computed tomography (CT) or magnetic resonance imaging (MRI).

SECONDARY OUTCOMES:
Eastern Cooperative Oncology Group (ECOG) evaluation | one to two years
  Complete an Eastern Cooperative Oncology Group (ECOG) evaluation
Haematology test | one to two years
  complete white blood cell count with differential, red blood cell count, hemoglobin, hematocrit, and platelets
Tumor marker measurement | one to two years
  measure the change of tumor marker such as carcinoembryonic antigen (CEA)
Conduct computed tomography (CT) or magnetic resonance imaging (MRI) scans for tumour response evaluation | one to two years
  Subjects will still be followed-up in the event of disease progression in order to document overall survival, a secondary endpoint.
Review concomitant medications | one to two years
  Use of medications will be reviewed and recorded
Assess for presence of adverse event | one to two years
  An adverse event assessment will be performed

CONTACTS AND LOCATIONS:
Overall Officials: Kai-Wen Huang, PhD, Principal Investigator — National Taiwan University Hospital

IPD SHARING:
Plan to Share IPD: No